CLINICAL TRIAL: NCT02972476
Title: Investigating the Mechanism of Inhaled Corticosteroids Associated Pneumonia by Longitudinal Characterisation of the Airway Microbiome in Patients With Severe COPD
Brief Title: Microbiome Use to Stratify Use of Inhaled Corticosteroids: MUSIC Trial
Acronym: MUSIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: AstraZeneca (Industry); NHS Tayside (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2014RC07; 2016-000734-21 (EudraCT Number)
Record Dates: First submitted 2016-10-18; First posted 2016-11-23 (Estimated); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide; Formoterol Fumarate; aclidinium bromide; Salmeterol Xinafoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1: Symbicort 400/12 & Eklira Genuair (Active Comparator): Budesonide 400mcg & formoterol fumarate 12mcg: 1 inhalation twice daily, inhalation powder and Aclidinium bromide 322mcg: 1 inhalation twice daily, inhalation powder for 3 months
  Interventions: Drug: Budesonide & formoterol fumarate and Aclidinium bromide
- 2: Seretide 500/50 & Eklira Genuair (Active Comparator): Fluticasone propionate 500mcg & salmeterol 50mcg: 1 inhalation twice daily, inhalation powder and Aclidinium bromide 322mcg: 1 inhalation twice daily, inhalation powder for 3 months
  Interventions: Drug: Fluticasone 500 & salmeterol and Aclidinium bromide
- 3: Seretide 250/50 & Eklira Genuair (Active Comparator): Fluticasone propionate 250mcg & salmeterol 50mcg: 1 inhalation twice daily, inhalation powder and Aclidinium bromide 322mcg: 1 inhalation twice daily, inhalation powder for 3 months
  Interventions: Drug: Fluticasone 250 & salmeterol and Aclidinium bromide
- 4: Duaklir Genuair (Active Comparator): Aclidinium bromide 340mcg & formoterol fumarate 12mcg: 1 inhalation twice daily, inhalation powder for 3 months
  Interventions: Drug: Aclidinium bromide & formoterol fumarate

INTERVENTIONS:
Drug: Budesonide & formoterol fumarate and Aclidinium bromide
  Other Names: Symbicort Turbohaler and Eklira Genuair
  Arms: 1: Symbicort 400/12 & Eklira Genuair
Drug: Fluticasone 500 & salmeterol and Aclidinium bromide
  Other Names: Seretide Accuhaler 500/50 and Eklira Genuair
  Arms: 2: Seretide 500/50 & Eklira Genuair
Drug: Fluticasone 250 & salmeterol and Aclidinium bromide
  Other Names: Seretide Accuhaler 250/50 and Eklira Genuair
  Arms: 3: Seretide 250/50 & Eklira Genuair
Drug: Aclidinium bromide & formoterol fumarate
  Other Names: Duaklir Genuair
  Arms: 4: Duaklir Genuair

SUMMARY:
A randomised controlled trial to test the hypothesis that inhaled therapies for chronic obstructive pulmonary disease (COPD) have differential effects on the upper airway microbiome.

COPD is the third leading cause of death worldwide. Exacerbations drive disease progression and worsening quality of life and therefore prevention of exacerbations has been a major goal of treatment.

Patients with COPD are frequently prescribed inhaled corticosteroids (ICS) which have been shown to reduce exacerbations in combination with long acting beta2-adrenoceptor agonists (LABA). In recent years, all ICS preparations have been associated with a significant increased risk of pneumonia in either randomised trials or observational studies leading to warnings from national regulatory authorities and leading experts. This has led to a re-evaluation of the role of ICS in COPD treatments. It is likely that the risk of pneumonia is not equal across all ICS doses and molecules.

There is a compelling rationale for ICS having a strong effect on the upper airway microbiome, and that this may be one mechanism of increased pneumonia risk with these drugs. The existing literature regarding ICS and pneumonia risk are lacking; 1) there are no head to head trials comparing different ICS preparations and 2) the comparator in these studies to date have been long acting beta2-adrenoceptor agonists alone, whereas the most appropriate comparator in current management would be combined LABA and long-acting muscarinic antagonist (LAMA).

The MUSIC TRIAL is a multi-centre randomised open label controlled parallel group study with four treatment arms and a total of 120 participants. Severe COPD patients currently treated with inhaled corticosteroid therapy will be randomised to treatment with one of three preparations of ICS in combination with LABA or the control arm of dual bronchodilator therapy following a four week washout period. Participants will return monthly to determine if there are changes in the microbiome in their upper airway.

This study will establish one potential mechanism for the increased susceptibility to pneumonia in ICS users and assess intraclass differences in ICS molecules and the effect of ICS dose on the microbiome. Demonstrating that different COPD treatments can have different effects on the lung microbiome is an important step in understanding clinical differences in the safety and effectiveness of different treatments for severe COPD.

DETAILED DESCRIPTION:
Inhaled corticosteroids (ICS) are commonly prescribed for patients with chronic obstructive pulmonary disease (COPD), but their role in the management of COPD is currently being re-evaluated in light of new evidence and the emergence of alternative treatments. Studies have shown that the use of ICS and particularly ICS combined with long acting beta2-adrenoceptor agonists (LABA) in individuals with COPD reduces the frequency of COPD exacerbations and improves health status and lung function compared to LABA alone or placebo. The current National Institute for Care Excellence (NICE) guidelines for COPD recommend ICS for patients with a forced expiratory volume in 1 second below 50% predicted, or for patients with higher lung function who have persisting symptoms or exacerbations despite treatment with long acting bronchodilators. Data suggests that up to 75% of patients with COPD in the United Kingdom (UK) are subsequently prescribed ICS.

The daily dose of ICS utilised in COPD treatments are much higher than those used in asthma treatments, with licensed daily doses being 1000 mcg fluticasone propionate (2000 mcg beclomethasone dipropionate (BDP) equivalents) or 800 mcg budesonide (800 mcg BDP equivalents).

Recent concerns have been expressed about the safety of ICS in COPD following several randomised controlled trials of fluticasone propionate and fluticasone furoate, among others, demonstrating an increase in rates of pneumonia as an adverse event. Several systematic reviews and observational studies confirm an association between ICS use and risk of pneumonia.

All ICS preparations have been associated with an increased risk of pneumonia in either randomised trials or observational studies leading to warnings from national regulatory authorities and leading experts.

It is likely however, that the risk of pneumonia is not equal across all ICS doses and molecules. Research into this area is greatly limited by the lack of head to head comparisons between different ICS preparations in COPD.

It is hypothesised that the anti-inflammatory and immunosuppressive effects of ICS lead to increase susceptibility to colonisation of the upper respiratory tract with pathogenic bacteria associated with pneumonia such as S. pneumoniae and Haemophilus influenzae. This study will establish one potential mechanism for the increased susceptibility to pneumonia in ICS users and assess intraclass differences in ICS molecules used in COPD and the effect of ICS dose. It is known that changes in the microbiome in COPD are associated with disease severity and with lung inflammation. Demonstrating that different COPD treatments can have different effects on the lung microbiome is an important step in understanding clinical differences in the safety and effectiveness of different treatments for severe COPD. The longer term clinical objective of this study is therefore to determine whether a proportion of patients with COPD might be more safely managed with either lower dose, pharmacologically different ICS preparations or with LABA/LAMA therapies to reduce the risk of pneumonia.

Hypothesis Fluticasone propionate will facilitate a higher level of bacterial airway colonisation by pathogens associated with pneumonia compared to budesonide or treatment exclusively with bronchodilators, therefore providing a mechanistic explanation for increased pneumonia risk associated with ICS.

STUDY OBJECTIVES To determine a potential mechanism of inhaled corticosteroid associated pneumonia in COPD by demonstrating ICS effects on the upper (throat and nasal swabs) and lower airway (sputum) microbiome.

To determine the mechanism of observed differences in pneumonia risk between fluticasone propionate, and budesonide by demonstrating differential effects on the airway microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged greater than or equal to 40 years
* Current or ex smokers having at least a 10 pack year smoking history
* A clinical diagnosis of Chronic Obstructive Pulmonary Disease (COPD) made by a physician with a post-bronchodilator forced expiratory volume 1 (FEV1)/ forced vital capacity (FVC) ratio at screening of <70%
* Severe COPD according to consensus guidelines consisting of a post-bronchodilator FEV1 <50% predicted at screening and/or a history of 2 or more exacerbations in the previous year OR one hospital admission for an exacerbation of COPD in the previous year (equivalent to Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2011 grade C and D)
* Able to perform all study procedures including spirometry and questionnaires with minimal assistance.

Exclusion Criteria:

* Inability to give informed consent
* Asthma (defined according to Scottish Intercollegiate Guidelines Network)
* A primary diagnosis of bronchiectasis confirmed on high-resolution computed tomography.(it is not necessary to perform a computerised tomography (CT) scan to exclude this if the patient has not previously had one. Only known bronchiectasis with a previous CT scan should be excluded).
* • Antibiotics within the past 28 days, apart from oral macrolides which are permitted if they have been used for at least 3 months prior to randomization
* Oral/ nasal corticosteroids of any kind in the 28 days prior to screening visit
* Current use of the following: roflumilast, ritonavir, itraconazole, telithromycin, or ketoconazole (or other CYP3A4 inhibitors).
* Active, or within 28 days of screening visit, oral candidiasis, actively receiving dental treatment for oral infection or poor dentition.
* Immunosuppression including current oral corticosteroids at a dose >5mg for >28 days.
* Glomerular filtration rate (eGFR) below 30ml/min/1.73meter squared or requiring dialysis. Last known eGFR result will be used .
* Use of any investigational drugs within five times of the elimination half-life after the last study dose or within 30 days, whichever is longer.
* Known allergy, intolerance or contraindication to any of the study drugs
* Galactose intolerance
* Unstable co-morbidities (cardiovascular disease, active malignancy) which in the opinion of the Investigator would make the patient unsuitable to be enrolled in the study. This includes any abnormality identified on screening bloods or screening electrocardiograph which in the opinion of the Investigator would make the patient unsuitable for the study.
* An exacerbation of COPD occurring during the screening to randomisation period. If this occurs the patient should be withdrawn from the study and may be rescreened once they have been free from corticosteroid and antibiotic treatment for 28 days. In these cases patients would receive the current Participant Information Sheet and be consented prior to starting the study from Visit 1.
* Documented that the patient has never received pneumococcal polysaccharide vaccination
* Receipt of Pneumococcal conjugate vaccine (e.g PCV-13)
* Pregnancy or breast feeding
* Women of child bearing potential (WOCBP) who are not practicing an acceptable method of contraception (see below)

Acceptable forms of contraception:

* combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, transdermal
* progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable, implantable
* intrauterine device (IUD)
* intrauterine hormone-releasing system ( IUS)
* bilateral tubal occlusion
* vasectomised partner
* sexual abstinence

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2016-12; Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
Change in bacterial load of total respiratory pathogens determined by quantitative polymerase chain reaction | Baseline, 1, 2, and 3 months
  To determine the effects of the inhaled corticosteroids fluticasone propionate/salmeterol 500/50 mcg vs budesonide/formoterol 400/12 mcg on upper airway bacterial load from oropharyngeal swabs.

SECONDARY OUTCOMES:
Change in bacterial load of total respiratory pathogens determined by quantitative polymerase chain reaction. | Baseline, 1, 2, and 3 months
  To determine the effects of the inhaled corticosteroids fluticasone propionate/salmeterol 500/50 mcg vs budesonide/formoterol 400/12 mcg on lower airway bacterial load and microbiome from sputum and on upper airway in nasophyarengeal swab.
Change in bacterial load of total respiratory pathogens determined by quantitative polymerase chain reaction. | Baseline, 1, 2, and 3 months
  To compare the effects of fluticasone/salmeterol 250/50mcg vs budesonide/formoterol 400/12 mcg on upper and lower airway microbiome in oropharyngeal/nasopharyngeal and sputum samples.
Microbiota diversity using the Shannon-Wiener diversity index determined by 16S microbiome sequencing | Baseline, 1, 2, and 3 months
  To determine the effects of the inhaled corticosteroids fluticasone propionate/salmeterol 500/50 mcg vs budesonide/formoterol 400/12 mcg on lower airway microbiome from sputum and on upper airway in nasopharyngeal swab. To compare the effects of fluticasone/salmeterol 250/50mcg vs budesonide/formoterol 400/12 mcg on upper and lower airway microbiome in oropharyngeal/nasopharyngeal and sputum samples.
Microbiota diversity using the Shannon-Wiener diversity index determined by 16S microbiome sequencing | Baseline, 1, 2, and 3 months
  To compare the effects of fluticasone/salmeterol 250/50mcg vs budesonide/formoterol 400/12 mcg on upper and lower airway microbiome in oropharyngeal/nasopharyngeal and sputum samples.
Microbiota diversity using the Shannon-Wiener diversity index determined by 16S microbiome sequencing | Baseline, 1, 2, and 3 months
  To compare the effects on the upper and lower airway microbiome in oropharyngeal, nasopharyngeal swabs and sputum of individual inhaled corticosteroids (ICS) fluticasone propionate and budesonide (pooled ICS group) compared to a dual bronchodilator based regime without ICS
Change in number of Operational Taxonomic Units of protocol defined respiratory pathogens. | Baseline, 1, 2 and 3 months
  To determine the effects of the inhaled corticosteroids fluticasone propionate/salmeterol 500/50 mcg vs budesonide/formoterol 400/12 mcg on lower airway microbiome from sputum and on upper airway in nasopharyngeal swab
Change in number of Operational Taxonomic Units of protocol defined respiratory pathogens. | Baseline, 1, 2 and 3 months
  To compare the effects of fluticasone/salmeterol 250/50mcg vs budesonide/formoterol 400/12 mcg on upper and lower airway microbiome in oropharyngeal/nasopharyngeal and sputum samples.
Change in number of Operational Taxonomic Units of protocol defined respiratory pathogens. | Baseline, 1, 2 and 3 months
  To compare the effects on the upper and lower airway microbiome in oropharyngeal, nasopharyngeal swabs and sputum of individual inhaled corticosteroids (ICS) fluticasone propionate and budesonide (pooled ICS) compared to a dual bronchodilator based regime without ICS
Change in airway microbiota bacterial species diversity measured using the Shannon Wiener diversity indexand beta diversity indices. | Baseline, 1, 2 and 3 months
  To compare the effects of fluticasone/salmeterol 250/50mcg vs budesonide/formoterol 400/12 mcg on upper and lower airway microbiome in oropharyngeal/nasopharyngeal and sputum samples.
Change in bacterial load of respiratory pathogens determined by quantitative polymerase chain reaction Microbiome characterisation | Baseline, 1, 2 and 3 months
  To compare the impact of high and low dose inhaled corticosteroid fluticasone propionate on the upper and lower airway microbiome in oropharyngeal, nasopharyngeal swabs and sputum
Change in bacterial load of respiratory pathogens determined by quantitative polymerase chain reaction | Baseline, 1, 2 and 3 months
  To compare the impact of high and low dose inhaled corticosteroid fluticasone propionate on the upper and lower airway microbiome in oropharyngeal, nasopharyngeal swabs and sputum
Changes in inflammatory markers in the sputum. | Baseline, 1, 2 and 3 months
  To evaluate the impact of inhaled corticosteroids on airway inflammation. Comparing inhaled corticosteroids to dual bronchodilator regimes alone. Measured with neutrophil elastase, myeloperoxidase, IL-8, IL-1beta.
Changes in inflammatory markers in the blood. | Baseline, 1, 2 and 3 months
  To evaluate the impact of inhaled corticosteroids on airway and systemic inflammation. Comparing inhaled corticosteroids to dual bronchodilator regimes alone. Measued with eosinophils & neutrophils, C-reactive protein, serum resistin, specific IgG antibody to bacterial pathogens.

OTHER OUTCOMES:
Comparison of adverse events/serious adverse events between groups on dual bronchodilators and inhaled corticosteroids | Baseline, 1, 2 and 3 months
  To evaluate the safety and tolerability of withdrawal of inhaled corticosteroids in severe Chronic Obstructive Pulmonary Disease
Change in Forced expiratory volume in 1 second | Baseline, 1, 2 and 3 months
  To evaluate the safety and tolerability of withdrawal of inhaled corticosteroids in severe Chronic Obstructive Pulmonary Disease
Change in patient self reported measures | Baseline, 1, 2 and 3 months
  To evaluate the safety and tolerability of withdrawal of inhaled corticosteroids in severe Chronic Obstructive Pulmonary Disease using St. George's Respiratory Questionnaire and Chronic Obstructive Pulmonary Disease Assessment Test score
Correlation between change in alpha and beta diversity indices and the frequency of adverse events | Baseline, 3 months
  To evaluate if changes in the airway microbiota are associated with AEs
Comparison of inflammatory markers before and after one month washout period. | -1 months and baseline
  To determine the impact of inhaled corticosteroids withdrawal on airway inflammation.
Comparison of bacterial load before and after one month washout period. | -1 months and baseline
  To determine the impact of inhaled corticosteroids withdrawal on airway bacterial load
Comparison of microbiome characterisation before and after one month washout period. | -1 months and baseline
  To determine the impact of inhaled corticosteroids withdrawal on airway microbiome.
Microbiota diversity determined by 16s microbiome sequencing using the Shannon Diversity index. | Baseline, 1, 2 and 3 months
  To provide a longitudinal characterisation of the upper and lower airway microbiome in oropharyngeal/nasopharyngeal swabs and sputum in Chronic Obstructive Pulmonary Disease
Bacterial community composition determined by 16s microbiome sequencing using number of reads of protocol defined respiratory pathogens. | Baseline, 1, 2 and 3 months
  To provide a longitudinal characterisation of the upper and lower airway microbiome in oropharyngeal/nasopharyngeal swabs and sputum in Chronic Obstructive Pulmonary Disease
Total bacterial load using qPCR | Start of decontamination period (washout) to end of decontamination period (baseline)
  To assess the effectiveness of chlorhexidine decontamination on lower airway microbiology in sputum in Chronic Obstructive Pulmonary Disease
Bacterial community composition determined by 16s microbiome sequencing | Start of decontamination period (washout) to end of decontamination period (baseline)
  To assess the effectiveness of chlorhexidine decontamination on upper and lower airway microbiology in Chronic Obstructive Pulmonary Disease
Bacterial community composition determined by 16s microbiome sequencing | Start of decontamination period (washout) to end of decontamination period (baseline)
  To assess the effectiveness of chlorhexidine decontamination on upper airway microbiome in sputum in Chronic Obstructive Pulmonary Disease
Quality of life- St Georges Respiratory Questionnaire | Baseline, 1 and 3 months
  To evaluate patient reported outcome measures on three different inhaled corticosteroids regimes compared to dual bronchodilator regimes using St. George's Respiratory Questionnaire and Chronic Obstructive Pulmonary Disease assessment test score
Comparison of oropharyngeal swabs with quantitative PCR, and 16s sequencing to measure validity, responsiveness and reliability comparing inhaled corticosteroids to dual bronchodilator regimes alone | Baseline, 1, 2 and 3 months
  To compare different microbiological methods for the assessment of changes in the upper and lower airway microbiome in COPD
Change in FEV1 | From baseline to 3 months follow-up.
  To evaluate if changes in the airway microbiome or airway inflammatory profiles are associated with efficacy or safety end-points
Comparison of time to first exacerbation of Chronic Obstructive Pulmonary Disease | From Baseline to 3 months
  To evaluate if changes in the airway microbiome or airway inflammatory profiles are associated with efficacy or safety end-points
Number of exacerbations of Chronic Obstructive Pulmonary Disease | Baseline, 3 months and as required, for example when an exacerbation occurs.
  To evaluate if changes in the airway microbiome or airway inflammatory profiles are associated with efficacy or safety end-points
Time to next exacerbation of Chronic Obstructive Pulmonary Disease | Baseline, 3 months and as required, for example when an exacerbation occurs.
  To evaluate if changes in the airway microbiome or airway inflammatory profiles are associated with efficacy or safety end-points

CONTACTS AND LOCATIONS:
Overall Officials: James Chalmers, MBChB, MRCP, Principal Investigator — University of Dundee
Locations (6):
- United Kingdom (6):
  - NHS Tayside, Dundee, Tayside
  - Blackpool Teaching Hospital NHS Foundation Trust, Blackpool
  - NHS Lothian, Edinburgh
  - NHS Greater Glasgow and Clyde, Glasgow
  - NHS Fife, Kirkcaldy
  - NHS Lanarkshire, Wishaw

IPD SHARING:
Plan to Share IPD: Undecided